CLINICAL TRIAL: NCT01850043
Title: The Trend of Tuberculin Skin Test in Korea
Brief Title: The Epidemiology of TST Change in Korea
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Assistant Professor, Asan Medical Center
Other Study IDs: KoreanTSTtrends
Record Dates: First submitted 2013-05-02; First posted 2013-05-09 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Tuberculosis; Latent Tuberculosis
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Military Conscripts: A term of whole military conscripts per year in one Reserve Force Battalion. Military conscripts gather from all around area in Korea randomly

SUMMARY:
TST will be analyzed in young general population in Korea. Young adults undertake TST as CDC recommendation. Participants with chest radiograph showing active TB lesion are excluded from this study.

DETAILED DESCRIPTION:
Enroll criteria

* A term of whole military conscripts per year in one Reserve Force Battalion
* Military conscripts gather from all around area in Korea randomly
* Each participant undertake a chest X-ray (CXR) and blood tests including human immunodeficiency virus (HIV) at the start of initiatory training.

Exclusion Criteria

* Chest X-ray suggesting active TB
* HIV positive in serology

Design

* After giving informed consent, all participants receive one-step TST following standard procedures.
* The largest transverse diameter of induration is measured 48-72hr after injection.
* The investigator and these trained nurses were blinded to the status of their demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Military Conscripts age 18-29 years old

Exclusion Criteria:

* Chest X-ray suggests active TB
* Positive HIV in serology

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A term of whole military conscripts per year
Sampling Method: Non-Probability Sample
Enrollment: 5552 (Actual)
Dates: Start 2005-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
TST positivity TST rate | Two days after tuberculin injection
  Investigators measure induration size of tuberculin skin test 48 after tuberculin injection.

SECONDARY OUTCOMES:
BCG scar rates | The day of tuberculin injection

CONTACTS AND LOCATIONS:
Overall Officials: HeeJin Kim, MD, Principal Investigator — The Korean Institute of Tuberculosis
Locations (1):
- The Korean Institute of Tuberculosis, Osong, North Chungcheong, South Korea